CLINICAL TRIAL: NCT05770531
Title: A Randomized Clinical Trial Comparing ctDNA-Directed Therapy Change With Standard of Care in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Circulating Tumor DNA to Guide Changes in Standard of Care Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vandana Abramson, Professor of Medicine, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICCBRE2257; NCI-2023-01721 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Metastatic HER2-Negative Breast Carcinoma; Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (biospecimen banking) (Active Comparator): Patients receive providers choice of standard of care chemotherapy and undergo blood sample collection for banking on study. Patients undergo CT or MRI during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Arm B (biospecimen evaluation, possible treatment change) (Experimental): Patients receive providers choice of standard of care chemotherapy and undergo blood sample collection for ctDNA evaluation on study. Patients may receive sacituzumab govitecan IV based on ctDNA results on study. Patients undergo CT or MRI during screening and on study.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Biological: Sacituzumab Govitecan

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection for banking
  Arms: Arm A (biospecimen banking)
Procedure: Computed Tomography — Undergo CT
Procedure: Magnetic Resonance Imaging — Undergo MRI
Procedure: Biospecimen Collection — Undergo blood sample collection for ctDNA evaluation
  Arms: Arm B (biospecimen evaluation, possible treatment change)
Biological: Sacituzumab Govitecan — Given by IV
  Arms: Arm B (biospecimen evaluation, possible treatment change)

SUMMARY:
This phase II trial tests how well evaluating circulating tumor deoxyribonucleic acid (ctDNA) works to guide therapy-change decisions in treating patients with triple-negative breast cancer (TNBC) that has spread from where it first started (primary site) to other places in the body (metastatic). This study wants to learn if small pieces of DNA associated with a tumor (called circulating tumor DNA, or ctDNA) can be detected in investigational blood tests during the course of standard chemotherapy treatment for breast cancer, and whether information from such investigational ctDNA blood testing could possibly be used as an early indication of chemotherapy treatment failure. It is hoped that additional information from investigational blood testing for ctDNA could help doctors to switch more quickly from a standard chemotherapy treatment that typically has significant side effects and which may not be working, to a different standard treatment regimen against TNBC, called sacituzumab govitecan. Sacituzumab govitecan is a monoclonal antibody, called hRS7, linked to a chemotherapy drug, called irinotecan. hRS7 is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as TROP2 receptors, and delivers irinotecan to kill them. Studying ctDNA may assist doctors to change therapy earlier if needed, and may improve health outcomes in patients with metastatic TNBC.

DETAILED DESCRIPTION:
Primary Objective:

- To determine whether patients with metastatic TNBC who undergo treatment changes guided by ctDNA dynamics demonstrate improved progression-free survival (PFS) compared to control patients assessed conventionally with imaging alone.

PRIMARY OBJECTIVE:

I. To determine whether patients with metastatic TNBC who undergo treatment changes guided by ctDNA dynamics demonstrate improved progression-free survival (PFS) compared to control patients assessed conventionally with imaging alone.

SECONDARY OBJECTIVES:

* To evaluate the overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in patients with metastatic TNBC who undergo treatment changes guided by ctDNA dynamics compared to control patients assessed by conventional imaging alone.
* To determine whether patients with metastatic TNBC who undergo treatment changes guided by ctDNA dynamics demonstrate improved PFS2 compared to control patients assessed with conventional imaging alone.
* To evaluate overall survival (OS) in patients with metastatic TNBC who undergo treatment changes guided by ctDNA dynamics compared to control patients assessed by conventional imaging alone.

EXPLORATORY OBJECTIVES:

* To evaluate for unique predictive values of ctDNA-defined clones identified through the blood-based analysis.
* To correlate ctDNA changes with standard imaging.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive providers choice of standard of care chemotherapy and undergo blood sample collection for banking on study.

ARM B: Patients receive providers choice of standard of care chemotherapy and undergo blood sample collection for ctDNA evaluation on study. Patients may receive sacituzumab govitecan intravenously (IV) based on ctDNA results on study.

Patients in both arms A and B undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and on study.

After completion of study treatment, patients are followed up at 3, 6, 9, and 12 months and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage IV (metastatic) estrogen receptor (ER), PR, HER2 negative invasive mammary carcinoma, previously documented by histological analysis and that meets the following criteria:

  * HER2 negativity is defined as any of the following by local laboratory assessment:

    * In-situ hybridization (ISH) non-amplified (ratio of HER2 to CEP17 < 2.0 or
    * Single probe average HER2 gene copy number < 4 signals/cell), or
    * Immunohistochemistry (IHC) 0 or IHC 1+ (if more than one test result is available and not all results meet the inclusion criterion definition, all results should be discussed with the sponsor-investigator to establish eligibility of the patient)
  * ER and PR negativity are defined as =< 10% of cells expressing hormonal receptors via IHC analysis
* PD-L1 negative (combined positive score [CPS] < 10) or otherwise not appropriate for checkpoint inhibitors
* Patients must have measurable disease according to the standard RECIST version 1.1

  * NOTE: CT scans or MRIs used to assess the measurable disease must have been completed with 28 days prior to the study drug initiation
* Patients must be age >= 18 years; both male and female are eligible
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study
* No prior chemotherapy regimens for metastatic disease
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained less than 28 days from initiation of study drug)
* Platelet count >= 100,000/mm^3 (obtained less than 28 days from initiation of study drug)
* Bilirubin, serum glutamic oxaloacetic transaminase (SGOT), serum glutatmic pyruvic transaminase (SGPT), alkaline phosphatase =< 4x upper limits of normal if no liver metastases present
* Serum total bilirubin must be < 3x upper limits of normal for patients with Gilbert disease
* Total bilirubin, SGOT, SGPT =< 6x upper limits of normal if liver metastases present (obtained less than 28 days from initiation of study drug)
* For patients who are not postmenopausal (women) or surgically sterile (absence of ovaries and/or uterus or vasectomy), agreement to remain abstinent or to use two adequate methods of contraception (e.g., condoms, diaphragm, vasectomy/vasectomized partner, tubal ligation), during the treatment period and for at least 30 days after the last dose of study treatment. Hormone based oral contraceptives are not allowed on study. Postmenopausal is defined as:

  * Age >= 55 years
  * Age =< 55 years and amenorrheic for 12 months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression; or follicle stimulating hormone and estradiol in the postmenopausal range

Exclusion Criteria:

* Leptomeningeal disease
* Uncontrolled tumor-related pain: patients requiring narcotic pain medication must be on a stable regimen at registration. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to randomization. Patients should be recovered from the effects of radiation. There is no required minimum recovery period. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not presently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to randomization
* Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > upper limit of normal [ULN]) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy
* Malignancies other than TNBC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biological therapy) other than the ones specified in the protocol
* Women only: pregnancy or lactation
* Evidence of significant uncontrolled concomitant disease that in the opinion of the investigator could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
* Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (class II or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina. Patients with a known left ventricular ejection fraction (LVEF) < 35% will be excluded. Patients with known coronary artery disease or congestive heart failure not meeting the above criteria must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
* Major surgical procedure within 4 weeks prior to randomization or anticipation of the need for a major surgical procedure during the course of the study other than for diagnosis. Placement of central venous access catheter(s) (e.g., port or similar) is not considered a major surgical procedure and is therefore permitted
* Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
  The study survival will be estimated using the Kaplan-Meier method with 95% confidence intervals (CIs). The CI based on the Greenwoods variance will be reported. In addition, the efficacy of the study groups will be compared for PFS with log-rank tests. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age, on the survival data. The adjusted p-values of the hazard ratios and the adjusted 95% confidence intervals will be reported.

SECONDARY OUTCOMES:
Incidence of adverse events | From initiation of study-indicated treatment until 30 days after final study-indicated treatment or until initiation of another anticancer therapy, whichever occurs first
  Adverse events will be graded according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events version 5.0. Adverse medical events will be tabulated. NCI toxicity grade 3 and grade 4 laboratory abnormalities will be listed.
Progression free survival 2 | Up to 3 years
  The study survival will be estimated using the Kaplan-Meier method with 95% CIs. The CI based on the Greenwoods variance will be reported. In addition, the efficacy of the study groups will be compared for PFS2 with log-rank tests. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age, on the survival data. The adjusted p-values of the hazard ratios and the adjusted 95% confidence intervals will be reported.
Overall survival (OS) | Up to 3 years
  The study survival will be estimated using the Kaplan-Meier method with 95% CIs. The CI based on the Greenwoods variance will be reported. In addition, the efficacy of the study groups will be compared for OS with log-rank tests. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age, on the survival data. The adjusted p-values of the hazard ratios and the adjusted 95% confidence intervals will be reported.
Response rate (RR) | Up to 3 years
  The exact two-sided 95% confidence intervals for the RR will be reported for each arm. The Fisher's exact test will be used to examine the difference of RR between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Abramson, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-06-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT05770531/ICF_000.pdf